CLINICAL TRIAL: NCT01844804
Title: Phase 1, Double Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Study of PF-06438179 and Infliximab Sourced From US and EU Administered to Healthy Volunteers
Brief Title: A Pharmacokinetics Study Comparing PF-06438179 and Infliximab in Healthy Volunteers (REFLECTIONS B537-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B5371001; REFLECTIONS B537-01
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Biosimilarity; Similarity; PK; Phase 1; Infliximab; Healthy Volunteers; Single-dose; Immunology
MeSH Terms: interventions — GP1111; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A = PF-06438179 (Experimental)
  Interventions: Biological: PF-06438179
- B = Infliximab-EU (Active Comparator)
  Interventions: Biological: Remicade
- C = Infliximab-US (Active Comparator)
  Interventions: Biological: Remicade

INTERVENTIONS:
Biological: PF-06438179 — Single-dose of 10 mg/kg administered as an intravenous infusion in not less than 2 hours on Day 1
  Other Names: Infliximab-Pfizer
  Arms: A = PF-06438179
Biological: Remicade — Single-dose of 10 mg/kg administered as an intravenous infusion in not less than 2 hours on Day 1
  Other Names: Infliximab (European Union)
  Arms: B = Infliximab-EU
Biological: Remicade — Single-dose of 10 mg/kg administered as an intravenous infusion in not less than 2 hours on Day 1
  Other Names: Infliximab (United States)
  Arms: C = Infliximab-US

SUMMARY:
In this study, healthy volunteers will receive a single intravenous dose of either PF-06438179 or infliximab (United States) or infliximab (European Union). During the course of the study, the pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms of PF-06438179 and the licensed infliximab products. Safety, tolerability, and immunologic response will also be evaluated throughout.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and healthy male subjects (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 32.0 kg/m2; and a total body weight >50kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant infectious, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, autoimmune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Previous exposure to a monoclonal antibody, or current use of other biologics.
* History of hypersensitivity reaction to inactive components of the study drugs or any murine proteins or anaphylactic reactions to therapeutic drugs.
* History of tuberculosis (TB) or a positive latent TB test at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Day 1 - Day 57
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUCt) | Day 1 - Day 57
Area Under the Curve From Time Zero Extrapolated to Infinite Time (AUCinf) | Day 1 - Day 57

SECONDARY OUTCOMES:
Systemic Clearance (CL) | Day 1 - Day 57
Terminal Disposition Half-Life (t1/2) | Day 1 - Day 57
Volume of Distribution at Steady State (Vss) | Day 1 - Day 57
Incidence of anti-infliximab antibodies (ADA), including neutralizing antibodies (Nab) | Day 1 - LSLV or Day 85 whichever occurs later

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Palaparthy R, Udata C, Hua SY, Yin D, Cai CH, Salts S, Rehman MI, McClellan J, Meng X. A randomized study comparing the pharmacokinetics of the potential biosimilar PF-06438179/GP1111 with Remicade(R) (infliximab) in healthy subjects (REFLECTIONS B537-01). Expert Rev Clin Immunol. 2018 Apr;14(4):329-336. doi: 10.1080/1744666X.2018.1446829. Epub 2018 Mar 12. PMID 29504427
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5371001&StudyName=A%20Pharmacokinetics%20Study%20Comparing%20PF-06438179%20and%20Infliximab%20in%20Healthy%20Volunteers%20%28REFLECTIONS%20B537-01%29